CLINICAL TRIAL: NCT03051113
Title: Identification of Neuromas by High Resolution Ultrasound in Patients With Peripheral Nerve Injury and Amputations
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: NeuromUL2016
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Neuropathic Pain; Neuroma
MeSH Terms: conditions — Neuralgia; Neuroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuromas are frequent after trauma and surgery, including amputation and can be identified by high-resolution ultrasound. The role of neuromas as the cause of neuropathic pain is uncertain. In this observational cohort study, the investigators wish to explore if the prevalence of neuromas are higher in patients with pain after peripheral nerve injury and amputation, than in patients with the same conditions but without pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with peripheral nerve injury 3 months prior to participation
* Subjects with amputation 3 months or more prior to participation

Exclusion Criteria:

* Severe somatic or psychiatric diseases
* Other peripheral neuropathy
* Lack of ability to cooperate to the clinical examination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral nerve injury after surgery or trauma. Amputees.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of neuromas in patients with pain and without pain after peripheral nerve injury or amputation. | 3 hours
  Neuromas identified by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Buch, MD, Principal Investigator — Department of Anesthesiology, Aarhus University Hospital
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No